CLINICAL TRIAL: NCT02797743
Title: Whole Blood Specimen Collection From Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progenity, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-111-HEALTHY
Record Dates: First submitted 2016-05-25; First posted 2016-06-13 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Whole blood from all ages and gender: - Ages from 0 to Adults (18 yrs of age or older)
  Interventions: Other: Whole blood

INTERVENTIONS:
Other: Whole blood — * Adults ≥18 yrs of age: up to 50 mL (5 tubes)
  * Adolescents 12-17 yrs of age: up to 30 mL (3 tubes)
  * Children 0-11 yrs of age: single tube (1 tube, 10 mL)

SUMMARY:
This study will obtain whole blood specimens from healthy subjects to be used for research and development and clinical validation of genetic assays.

DETAILED DESCRIPTION:
Progenity is developing diagnostic products to improve the healthcare of men, women, and children. The commercial objective is to make safe, noninvasive genetic testing available to the public, independent of age and other factors that may contribute to pregnancy or other clinical complications.

Sample specimens will not be used to develop genetic lines and/or DNA banks for cloning. Any samples or remnant specimens remaining may be stored indefinitely for future research programs.

Eligible subjects (or parent/guardian) will provide written informed consent after which basic demographic and clinical data will be obtained and a whole blood sample will be collected. A subject's participation may end immediately after their blood draw. The amount of whole blood drawn at any visit will be based upon age of the subject and test to be performed.

In the event a Subject is pregnant, information regarding the gender of the fetus established by either ultrasound, non-invasive prenatal testing (NIPT) results, or at delivery will be collected. Clinical data regarding any karyotyping procedure that may occur on the fetus will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or guardian)is willing to provide written informed consent to have up to 50 mL of whole blood collected at a single clinic visit (maximum blood volume will depend on age of subject)
* Subject is considered healthy (and if pregnant, their pregnancy is progressing normally)
* If pregnant, Subject is carrying a singleton fetus of 10 to 26 weeks' gestational age inclusive

Exclusion Criteria:

* Women who are not pregnant
* If pregnant, pregnancy is non-viable
* If pregnant, evidence of or suspected fetal anomaly based on ultrasound finding, abnormal 1st trimester screening or abnormal NIPT
* Immediate family history of a previous fetal aneuploidy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Men, pregnant women or children, no age restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Whole blood collection | about 3 years
  Whole blood collection from 750 healthy subjects total

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stiegler, PhD, Study Director — Head of Clinical Affairs
Locations (3):
- United States (3):
  - Heinen Obstetrics & Gynecology, Eunice, Louisiana
  - Virtua Medical Group, Voorhees Township, New Jersey
  - Cincinnati Obgyn, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No